CLINICAL TRIAL: NCT05662293
Title: Arrhythmia-induced Cardiomyopathy - a Prospective Observational Cohort Study
Brief Title: Characterization of Arrhythmia-induced Cardiomyopathy
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-00873; kt22Badertscher2
Record Dates: First submitted 2022-12-14; First posted 2022-12-22 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Cardiomyopathy; Arrhythmia-induced Cardiomyopathy (AiCM)
Keywords: atrial fibrillation (AF); supraventricular tachycardia (SVT); ventricular tachycardia; atrial flutter; Major Adverse Cardiovascular Event (MACE); cardiac arrhythmia
MeSH Terms: conditions — Cardiomyopathies; Atrial Fibrillation; Tachycardia, Supraventricular; Tachycardia, Ventricular; Atrial Flutter; Arrhythmias, Cardiac | interventions — omega-Chloroacetophenone; Quality of Life; Surveys and Questionnaires; Data Collection; Retrospective Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with arrhythmia-induced cardiomyopathy (retrospective/prospective): retrospective cohort and case-control study followed by a prospective observational cohort study.
  Interventions: Other: Data collection: Major adverse cardiovascular event (MACE) assessment questionnaire (prospective part); Other: Data collection: Quality of Life (QoL) Questionnaire (prospective part); Other: Data collection (retrospective study); Other: Data collection (prospective study database)

INTERVENTIONS:
Other: Data collection: Major adverse cardiovascular event (MACE) assessment questionnaire (prospective part) — Data collection: Major adverse cardiovascular event (MACE) assessment questionnaire (prospective part). The assessment will be done via mail, letter or phone
Other: Data collection: Quality of Life (QoL) Questionnaire (prospective part) — Data collection: Quality of Life (QoL) Questionnaire (prospective part). The questionnaire "EQ-5D-5L questionnaire" will be used to assess quality of life.
Other: Data collection (retrospective study) — Anonymized search and review of patients electronic health records of the University Hospital of Basel for patients with a reduced LVEF and a concomitant (±1year or after any observation of a reduced LVEF in imaging) diagnosis of arrhythmia known to be causing AiCM.
Other: Data collection (prospective study database) — Data collection on alcohol consumption, family history, rhythm disorder, hospitalizations, cardiac assessments, adverse events at baseline, 6 months, 1 year, 2 years and 5 years.

SUMMARY:
The goal of the this observational study is to gather clinically available data on patients presenting with a suspicion for arrhythmia-induced cardiomyopathy (AiCM) at the University Hospital Basel.

DETAILED DESCRIPTION:
Current studies indicate that AiCM is an under-recognized and an underestimated clinical entity and its prevalence is poorly documented. This project consists of a retrospective longitudinal cohort and case-control study followed by a prospective observational cohort study.

The retrospective pilot study (1200 patients) is to define the incidence of AiCM in patients who presented to the University Hospital of Basel with a reduced left ventricular ejection fraction before or after the diagnosis of an arrhythmia suggestive to lead to an AiCM.

The prospective study part (1500 patients) is to evaluate the predictors of adverse events and re-hospitalizations in patients with a suspicion of AiCM. The diagnosis of AiCM will be established using a "goldstandard diagnosis": 2 independent cardiologists will adjudicate the diagnosis based on all data from the initial hospital stay and follow-up including ECG, laboratory measurements, vital signs, echocardiography, coronary angiography, stress testing and other cardiovascular diagnostic steps. The most likely diagnosis will be chosen among a list of comprehensive, pre-selected choices. In cases of disagreement of the two reviewers, diagnosis will be discussed with a third senior physician and decision made.

In order to optimize the care of patients with AiCM, the researchers intend to determine the prevalence of AICM, evaluate diagnostic criteria that allow an early diagnosis of AICM, and evaluate the current therapeutic management and prognosis of patients with AICM.

ELIGIBILITY:
Prospective part

Inclusion Criteria:

* Diagnostic or suspicion of AiCM as presence of specified keyword in patient's file or as screened by colleagues of the internal medicine or cardiology clinics
* Signed study consent

Exclusion Criteria:

* Patient's active refusal of the general consent of the University Hospital Basel
* Age <18 years old
* Temporary exclusion criteria: Acute health condition such as myocardial infarction, patients presenting with a major trauma, a sepsis, patients shortly after cardiac surgery, and patients in shock (>100 bpm, <90 systolic BP, evidence of organ dysfunction).
* Life expectancy <1 year (palliative, terminal cancer)

Retrospective part

Inclusion Criteria:

* Patients with a reduced left-ventricular ejection fraction (LVEF ≤50%) or a reduction of 15% in the ejection fraction (EF) between two echocardiographies and a concomitant diagnosis of any arrhythmia likely to lead to AiCM within one year before or after diagnosis of the reduced LVEF from 2010-2021

Exclusion Criteria:

* Age < 18 years old
* Patient's active refusal of the general consent of the University Hospital Basel
* Acute event clearly leading to an acutely reduced LVEF (massive type I myocardial infarction, cardiogenic shock from a coronary or myocardial etiology, septic shock leading to toxic myopathy, hypovolemic shock with reduced EF, cardiac arrest and/or need for resuscitation).
* Patients with life expectancy <1 year (palliative, terminal cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective part (1500 patients):
  Patients which have been or currently are in treatment for an AiCM at the University Hospital Basel or who received a new diagnosis/suspicion of such a disease will be included. Patients who have just recovered from an AiCM they presented in the last 10 years will also be enrolled and prospectively followed.
  Retrospective part (1200 patients):
  Patients with a reduced LVEF (≤50%) or with a reduction of the EF of 15% between two echocardiographies and a concomitant diagnosis of arrhythmia (within one year prior or after the diagnosis of reduced EF) at the University Hospital Basel will be retrospectively identified by conducting a search in the electronic records for keywords of arrhythmia diagnosis and/or reduced EF in several imaging types.
Sampling Method: Probability Sample
Enrollment: 2700 (Estimated)
Dates: Start 2021-06-10 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of AiCM (retrospective part of the study) | one time data extraction and analysis at baseline
  Categorization (based on a diagnostic algorithm) into 4 categories: "Likely AiCM", "possibly AiCM", "unlikely AiCM" and "Diagnostic work-up and longitudinal assessment insufficient to establish diagnosis" done by study team. AiCM will be defined as the presence of a reduced (<50%) ejection fraction in a transthoracic echocardiography (TTE) with a concomitant diagnosis of an arrhythmia present in the electronic patient's chart 6 months before or after the date of the diagnostic study.
Incidence of AiCM (Prospective part of the study) | at 1 year Follow- up
  Categorization using a "goldstandard diagnosis (GSD)": diagnosis by 2 independent cardiologists based on all data from the initial hospital stay and follow-up. The most likely diagnosis will be chosen among a list of comprehensive, pre-selected choices (Standard operating procedures (SOP) provided to the adjudicators to ensure homogenous knowledge and adjudication process. The booklet will contain information from the guidelines and position papers)
Change in Major adverse cardiovascular events (MACE) assessment questionnaire | at 6 months, 1 year, 2 year and 5 year Follow- up
  MACE is a composite endpoint of nonfatal stroke, nonfatal myocardial infarction, and cardiovascular death.

SECONDARY OUTCOMES:
Percentage of patients in whom a diagnosis of AiCM could be diagnosed or excluded with certainty per goldstandard diagnosis. (prospective part) | up to 5 years
  Data generated by patient's chart review and automated IT export
Percentage of patients in whom a diagnosis of AiCM could not surely be established and/or where an overlap with another cause of cardiomyopathy was present per goldstandard diagnosis. (prospective part) | up to 5 years
  Data generated by patient's chart review and automated IT export
Percentage of patients in whom the goldstandard diagnosis procedures came to a different diagnosis than the one done by the clinician. (prospective part) | up to 5 years
  Data generated by patient's chart review and automated IT export
Frequency of hybrid (both antiarrhythmics and ablation) or a sequential (first anti-arrhythmic and then ablation) therapeutic options (prospective part) | one time data extraction and analysis
  Data generated by patient's chart review and automated IT export
Number of patients with tachymyopathies (prospective part) | up to 5 years
  supraventricular tachycardias such as atrial fibrillation, atrial flutter or atrial tachycardia vs premature-ventricular complex induced arrhythmia-induced cardiomyopathy versus right-ventricle pacing induced arrhythmia-induced cardiomyopathy
Change in European Quality of Life 5 Dimensions (EQ-5D-5L) quality of life (QoL) questionnaire in patients with and without a arrhythmia-induced cardiomyopathy (prospective part) | at 6 months, 1 year, 2 year and 5 year Follow- up
  The EQ-5D-5L consists of 2 parts: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels. The patient is asked to indicate his/her health state by ticking the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Badertscher, MD, Principal Investigator — University Hospital Basel, Department of Cardiology
Locations (1):
- University Hospital Basel, Department of Cardiology, Basel, Switzerland